CLINICAL TRIAL: NCT05636384
Title: SupporTive Care At Home Research (STAHR): a Cluster Non-randomized Controlled Trial for Patients With Advanced Cancer
Brief Title: SupporTive Care At Home Research for Patients With Advanced Cancer (STAHR-cancer)
Acronym: HOMECARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); DongGuk University (Other); Kyung Hee University Hospital (Other); Bundang CHA Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BeLong Cho, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HC21C0115-1
Record Dates: First submitted 2022-10-17; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Malignant Neoplasm; Home Care Services; Quality of LIfe; Unplanned Hospitalization
MeSH Terms: conditions — Neoplasms | interventions — Home Care Services, Hospital-Based

STUDY DESIGN:
Intervention Model Description: A cluster, non-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients enrolled in the intervention cluster (institution) are given specialized home-based medical care based on a specialized home-based medical team approach.
  Interventions: Other: Home-based care
- Control (No Intervention): Patients enrolled in the control cluster (institution) are only given the educational materials.
  Except for the home-based care intervention, usual care for advanced cancer patients was not restricted for these patients.

INTERVENTIONS:
Other: Home-based care — Home-based medical care is based on a specialized home-based medical team approach, including following:
  1. Specialized Home-Based Medical Team Approach
  2. Initial Assessment and Education
  3. Initial Home Visits and Education
  4. Multidisciplinary Team Meeting
  5. Regular Assessment After the Initial Visit
  Arms: Intervention

SUMMARY:
To test the effects of home-based care on unplanned hospitalization within 6 months among advanced cancer patients with decreased performance status. Home-based care includes education for patients and their family caregivers, home visits by specialized home-based medical staff, and regular status check-ups.

DETAILED DESCRIPTION:
This study is a cluster, non-randomized controlled trial to test the effects of home-based care on unplanned hospitalization in 6 months among advanced cancer patients with decreased performance status. Home-based care includes education for patients and their family caregivers, home visits by specialized home-based medical staff, and regular status check-up. We are recruiting the study participants from 6 institutions, aiming for 396 cancer patients.

Participants for the intervention group will be recruited from Seoul National University Hospital, Chung-ang University Hospital, and Dongguk University Ilsan Hospital. Participants for the control group will be recruited from Kyung Hee University Medical Center, CHA Bundang Medical Center, and Seoul National University Bundang Hospital.

ELIGIBILITY:
Inclusion Criteria:

Both the patient and their family caregiver must meet the criteria to be considered for this research.

1. Patient

   1. A person who has an advanced-stage solid cancer diagnosis (ICD-10 code C00-C70); A person who is receiving or planning to receive cancer treatment
   2. A person who meets one of the following conditions

      1. Has been evaluated as having ECOG performance status 2
      2. Has been evaluated as having ECOG performance status 1 and is over 70 years of age
   3. A person who wishes to stay at home
   4. A person whose family caregiver resides at home
   5. A person who wishes to participate in the research
2. Family Caregiver

   1. A family* member of the patient

      * Family: refers to the patient's spouse (including a common-law partner), descendants and their spouses up to the second degree, siblings and their spouses, and relatives and their spouses up to the eighth degree.
   2. A person who meets one of the following conditions:

      1. Lives with the patient (patient's household member)
      2. Does not live with the patient, but visits the patient's home more than three times a week
   3. A person who wants the patient to stay at home
   4. A person who can communicate easily with medical staff
   5. A person who wishes to participate in the research

Exclusion Criteria:

If either the patient or the family caregiver meets any one of these criteria, they are excluded from the study.

1. Patient

   1. A person who cannot speak, hear, or read Korean
   2. A person who is judged by a medical doctor to be unable to take part in this research due to extremely poor health
   3. A person residing outside the range that can be visited by the respective medical institution (the conditions for distance are to be specified by each medical institution)*

      * This condition is not applicable for the control group.
   4. A person who has used hospital- or home-type hospice and palliative care services
   5. A person who is under the age of 19
2. Family Caregiver

   1. A person who cannot speak, hear, or read Korean
   2. A person who is judged by a medical doctor to be unable to take part in this research due to extremely poor health
   3. A person under the age of 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospitalization | within 6 months following enrollment
  1. admission to the enrolled hospital to treat unexpected symptoms or medical conditions (not including planned admission for chemotherapy or admission for planned surgery or intervention)
  2. admission to a hospital other than the enrolled hospital
  3. admission to a nursing hospital for a duration of less than 4 weeks.

SECONDARY OUTCOMES:
Patient medical utilization | within 6 months following enrollment
  The total number of hospital utilization, including hospitalization, emergency room visit, and clinic visits
Hospitalization | within 6 months following enrollment
  the number of hospitalization
ER visits | within 6 months following enrollment
  the number of emergency room visits
Healthcare use | within 6 months following enrollment
  the number of healthcare use for severe diseases
Patient end-of-life care: ICU admission | within 1 month before death
  ICU admission one month before death
Patient end-of-life care: ventilator treatment | within 1 month before death
  Mechanical ventilator apply one month before death
Patient end-of-life care: an advance directive | within 1 month before death
  Completion of advance medical directives within 1 month before death
Quality of life of patient - ESAS | within 6 months following enrollment
  Modified Edmonton Symptom Assessment System (ESAS) of patient
Quality of life of patient - EQ-5D | within 6 months following enrollment
  Euro-Quality of Life-5 Dimension (EQ-5D) of patient
Depressive symptom of patient | within 6 months following enrollment
  Patient Health Questionnaire-9 (PHQ-9) of patient
Satisfaction with services (patient) | within 6 months following enrollment
  Satisfaction of the study participant (patient) with the service in this study, evaluated by questionnaire
Quality of life of family caregiver | within 6 months following enrollment
  Euro-Quality of Life-5 Dimension (EQ-5D) of family caregiver
Care burden of family caregiver | within 6 months following enrollment
  The Korean version of Caregiver Reaction Assessment (CRA-K) of family caregiver
Depressive symptom of family caregiver | within 6 months following enrollment
  Patient Health Questionnaire-9 (PHQ-9) of family caregiver
Caring competency of family caregiver | within 6 months following enrollment
  Caring competency of family caregiver, measured by questionnaire
Satisfaction with services (family caregiver) | within 6 months following enrollment
  Satisfaction of the study participant (family caregiver) with the service in this study, evaluated by questionnaire
Expenses | within 6 months following enrollment
  medical expenses, care expenses

CONTACTS AND LOCATIONS:
Overall Officials: Belong Cho, MD, MPH, PhD, Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Dongguk University Medical Center, Goyang-si, Gyeonggi-do
  - Bundang CHA Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Chung-Ang University Hosptial, Seoul
  - Kyung Hee University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No